CLINICAL TRIAL: NCT02431715
Title: [18 F]-6-L-fluorodihydroxyphenylalanine (18F-FDOPA) Positron Emission Tomography (PET) in Neuroendocrine Tumours
Brief Title: 18F-FDOPA PET in Neuroendocrine Tumours
Status: No longer available | Type: Expanded Access
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H12-01795
Record Dates: First submitted 2015-04-27; First posted 2015-05-01 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2022-11

CONDITIONS: Thyroid Cancer, Medullary; Carcinoid Tumor; Pheochromocytoma; Paraganglioma; Insulinoma; Neuroblastoma
MeSH Terms: conditions — Thyroid cancer, medullary; Carcinoid Tumor; Pheochromocytoma; Paraganglioma; Insulinoma; Neuroblastoma | interventions — fluorodopa F 18

INTERVENTIONS:
Drug: [18 F]-6-L-fluorodihydroxyphenylalanine (18F-FDOPA) — All patients will have their weight and baseline vital signs recorded.
  The study subject will have an intravenous catheter inserted and receive a slow bolus intravenous dose of 185 - 370 MBq (5 -10mCi) 18F-FDOPA.
  The patient will rest in a comfortable reclining chair in a warm, private shielded room for 45 to 60 minutes.
  Patients are positioned supine and centered on the scanner bed for an average total scan time (CT and PET) of approximately 30 minutes.
  Images will be interpreted by qualified and experienced physicians. Findings of significance from the PET/CT scan, and any incidental findings of significance from the CT scan, will be included in the single final report that will be issued to referring physicians.
  Other Names: 18F-FDOPA

SUMMARY:
Neuroendocrine tumours (NETs) are a group of neoplasms generally arising from the gastroenteropancreatic tract. They are usually slow growing, have low malignant potential, and often go unnoticed until they become metastatic. The correct treatment approach is dependent on the extent of the disease, however surgical approaches and systemic therapy can be curative.

Combined positron emission tomography/computed tomography (PET/CT) using the radiotracer 18F-6-L-fluorodihydroxyphenylalanine (18F-FDOPA) has been shown to be a promising non-invasive technique to help localizing NETs and guide their treatment.

DETAILED DESCRIPTION:
Purpose/Objective:

The purpose of this study is to provide access to 18F-6-L fluorodihydroxyphenylalanine (18F-FDOPA) positron emission tomography and computed tomography (PET/CT) imaging to patients with neuroendocrine tumours (NET) and to collect additional data about the effectiveness of 18F-DOPA PET/CT in this patient population.

Hypothesis:

1. The overall accuracy of 18F-FDOPA PET/CT is superior to conventional imaging techniques for the detection of neuroendocrine tumours.
2. The sensitivity of 18F-FDOPA PET/CT is superior to conventional imaging techniques for the detection of neuroendocrine tumours.

Justification:

Treatment of NET's depends on the extent of disease and rate of tumour progression. Accurate staging is critical to establish the prognosis of the disease, to guide potentially curative surgical approaches and to assist in therapeutic decision making between surgery, embolization techniques and systemic therapy. Standard radiologic and nuclear medicine techniques all have significant limitations in terms of their ability to detect these lesions and to evaluate response to treatment. The widely used PET tracer 18F-Fluorodeoxyglucose (18-FDG) is of limited value in NET's due to its non-specific uptake and the relatively low mitotic rate often seen in these tumours.

Combined PET/CTutilizing 18F-FDOPA has been investigated as a potentially sensitive and specific staging and localization technique for NETs. Expression of tumour-specific catecholamine transport and storage mechanisms by NET cells is the basis of 18F-DOPA PET imaging. Cellular uptake and radiopharmaceutical concentration in intracellular storage granules within tumour cells of neuroendocrine origin and differentiation, combined with the high sensitivity, resolution and accurate anatomic localization of PET/CT imaging, makes 18F-DOPA PET/CT potentially superior to standard nuclear medicine and radiologic techniques for the detection and localization of functioning and non-functioning NETs. This imaging technique not only provides specific functional and biochemical information via PET images, but also morphological and anatomical detail via CT images leading to more accurate localization and characterization on individual lesions. This may allow better treatment planning as well as restaging during and after therapy to assess disease response. The information retrieved from the hybrid 18F-FDOPA PET/CT could have a profound influence on diagnosis and treatment of patients with NETs.

Research Method:

This will be an expanded access study in which adult and pediatric subjects will be invited to participate. All subjects are informed of anticipated effects (none) and purpose of the injected substance. Subjects are approached by their treating physicians with respect to their willingness to participate in the proposed study based on clinical criteria. They will then undergo a brief clinical assessment followed by the PET/CT scanning protocol.

The BC Cancer Agency anticipates a start date in August 2012 and a potential completion date August of 2017. Three full years of data collection will provide meaningful numbers for analysis. A total of 300 patients, including adults and pediatric patients, will be recruited for the study. This number is based on the anticipated number of PET scan referrals expected over a five-year study timeframe.

Statistical Analysis:

The primary outcomes will be estimates of sensitivity, specificity and accuracy of 18F-DOPA PET. 95% confidence intervals will be calculated for all estimates. Outcomes will be estimated for the whole study population and for different types of cancer.

Sensitivity (ratio of true positive lesions to total positive lesions), specificity (ratio of true negative lesions to total negative lesions) and accuracy (ratio of total correct studies to the total number of biopsied lesions) of 18F-FDOPA PET studies performed by the BCCA will be obtained by comparing results of the PET scan with the gold-standard of histopathological diagnosis when those results are available (as determined by clinical indication and feasibility by the treating physician) and results of conventional imaging. Biopsy of lesions is not mandated by this study. Confidence intervals (95% CI) for sensitivity, specificity and accuracy will be calculated using exact binomial distribution.

Results will be compared to figures in the published literature. All analyses will be performed in direct consultation with a statistician who is a member of the BC Cancer Agency staff.

ELIGIBILITY:
Inclusion Criteria

* Patients who meet the BCCA approved clinical indications for 18F-FDOPA PET/CT scans in neuroendocrine tumours.
* ECOG performance status 0 - 3.
* Able to provide written informed consent (or consent by guardian for subjects <19 years).
* Referred by a treating BC physician.
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 40 minutes and tolerating intravenous cannulation for injection.

Exclusion Criteria

* Pregnancy.
* Patients who are medically unstable eg. acute cardiac or respiratory distress, hypotensive
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70 cm).

Min Age: 1 Month | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada